CLINICAL TRIAL: NCT05413395
Title: Assessment of the Effects on the Skin Microbiome of Amending an Over-the-counter Eczema Product With Activated Oil (AO)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GlycosBio, Inc. (Industry)
Collaborators: Center for Clinical Studies, Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLYCOS-002-AD22
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, blinded, controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protocol (Experimental): Standard-of-care (SOC), over-the-counter (OTC) topical colloidal oatmeal formulation with a modified plant oil ("Activated Oil", AO) applied to designated "target lesion sites" and "non-lesion sites" (study sites) twice per day for 14 days, followed by a 7-day regression durability period during when no product is applied.
  Interventions: Other: topical colloidal oatmeal formulation with a modified plant oil
- Control (Active Comparator): Standard-of-care (SOC), over-the-counter (OTC) topical colloidal oatmeal formulation amended with deionized water to match the colloidal oatmeal concentration of the Protocol arm applied to designated "target lesion sites" and "non-lesion sites" (study sites) twice per day for 14 days, followed by a 7-day regression durability period during when no product is applied.
  Interventions: Other: topical colloidal oatmeal formulation

INTERVENTIONS:
Other: topical colloidal oatmeal formulation with a modified plant oil — Standard-of-care (SOC), over-the-counter (OTC) topical colloidal oatmeal formulation with a modified plant oil ("Activated Oil", AO). The AO contains proprietary blends of plant oils that have selective antimicrobial properties.
  Arms: Protocol
Other: topical colloidal oatmeal formulation — Standard-of-care (SOC), over-the-counter (OTC) topical colloidal oatmeal formulation
  Arms: Control

SUMMARY:
This is a single-center, randomized, blinded, controlled trial assessing the effects on the skin microbiome in patients with eczema of amending a standard-of-care (SOC), over-the-counter (OTC) topical colloidal oatmeal formulation with a modified plant oil ("Activated Oil", AO)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female subjects aged who have a recent eczema itch flareup and/or pre-flare-up symptoms at screening as determined by visual analog scale (VAS).
* Diagnosis of mild to moderate eczema (grade 3 - 7 on the Rajka-Langeland severity index).
* Having a target lesion with an ADSI score of 6-12 and an erythema and pruritus subscore of ³2 (moderate).
* Generally good health based on reported history.
* Able to discontinue all medical and over the counter topical emollients, moisturizers, and / or other skin barrier lotions.
* Females of child-bearing potential should agree to continue using a medically acceptable method of birth control throughout the study and for 30 days immediately after the last dose of study drug.
* Ability to administer topical medication and be willing to adhere to the study interventions.
* Agreement to adhere to Lifestyle Considerations throughout the duration of the study.

Exclusion Criteria:

* Pregnancy or lactation.
* Any type of malignancy involving the Study Site Area (Lesion or Non-Lesion site) in the last 5 years.
* Known allergy to hydrocortisone or topical antibiotic.
* Topical or oral use of an antibiotic within the last 7 days prior to baseline clinical visit.
* Bleach bathing in the 7 days prior to Baseline clinical visit.
* Current use of Class I-III topical corticosteroids or systemic medications (e.g. Dupixent) potentially affecting eczema or the skin.
* Surgeries or invasive medical procedures planned during course of study.
* Suspected non-compliance or non-cooperation.
* Intake of experimental drugs or experimental topical skin treatments within 30 days prior to study start.
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subject's participation in or ability to complete the study.
* Diagnosis of human immunodeficiency virus in medical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Atopic Dermatitis Severity Index (ADSI) score | 14 days
  Change in mean Atopic Dermatitis Severity Index (ADSI) score from baseline between the protocol and control arms by the 14-day application period. The ADSI comprises an assessment of erythema, pruritus, exudation, excoriation, and lichenification, each on a scale of 0 to 3 to give a maximum score of 15. The maximum score means a worsen condition.
Change in absolute abundance of S. aureus on target lesion site | 14 days
  Difference in reduction in absolute abundance of S. aureus on target lesion site compared to initial absolute abundance at target lesion site (Baseline measurement) between the protocol and control arms by 14-day application period of application period.

SECONDARY OUTCOMES:
Change in relative abundance of S. aureus on non-lesion site | 14 days
  Change in relative abundance of S. aureus on non-lesion site compared to initial relative abundance at target lesion site (Baseline measurement) between the protocol and control arms.
Change in absolute abundance of S. aureus and S. epidermidis on target lesion versus non-lesion site. | 14 days
  Change in absolute abundance of S. aureus and S. epidermidis on the target lesion site compared to the initial absolute abundance of S. aureus and S. epidermidis at the non-lesion site (Baseline measurement) between the protocol and control arms.
Change in Shannon Diversity Index between the target lesion site and non-lesion site | 14 days
  Change in Shannon Diversity Index between the target lesion site compared to the initial Shannon Diversity Index at the non-lesion site (Baseline measurement).
Change in Eczema Area and Severity Index (EASI) score | 14 days
  Change in mean Eczema Area and Severity Index (EASI) score from baseline between the protocol and control arms. An EASI score is a tool used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). For more information, see Hanifin JM, et al. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Studies, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No